CLINICAL TRIAL: NCT01333202
Title: Efficacy of Fresh Lime Alone for Smoking Cessation
Brief Title: Fresh Lime Alone for Smoking Cessation
Acronym: LIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Health Professional Alliance Against Tobacco (Other)
Responsible Party: Dr.Suthat Rungruanghiranya, Faculty of Medicine, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50-00-0980-02/2552
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2010-08

CONDITIONS: Tobacco Use Disorder
Keywords: Fresh lime; nicotine gum; smoking cessation; craving
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — lime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh lime (Experimental): Those who were randomly assigned to receive fresh lime were instructed to use it every time they began to crave cigarettes and as often as they needed. Fresh lime needed to be washed and cut into several small pieces by 1st cutting each lime into quarters and then each quarter further into 4 pieces. When needed, subjects were told to suck each piece of lime and thereafter chew the lime skin. To maintain freshness, the remaining slices were to be covered with plastic wrap and stored in the refrigerator as soon as possible. All participants in this group had to report the number of fresh lime slices used per day in the self-report card.
  Interventions: Other: Fresh lime
- Nicotine gum (Active Comparator): The dosage of nicotine gum used in this group was primarily based on the participants' FTND scores. Those with FTND score of 4 or above were given 4-mg nicotine gum. The 2-mg gum was assigned only to light smokers. Appropriate gum use by "chew and park" technique was instructed to all subjects in this group. They were advised to use the gum whenever they began to crave a cigarette but not to exceed more than 20 pieces per day. All participants in this group also had to report the total number pieces of gum used per day in the self-report card. Like the lime use group, phone calls were also made every 2-3 days during the initial month of study to remind them of technique and record keeping.
  Interventions: Other: Fresh lime

INTERVENTIONS:
Other: Fresh lime — fresh lime were used every time the participants began to crave cigarettes and as often as they needed. To correctly use it, fresh lime needed to be washed and cut into several small pieces by 1st cutting each lime into quarters and then each quarter further into 4 pieces. When needed, subjects were told to suck each piece of lime and thereafter chew the lime skin. To maintain freshness, the remaining slices were to be covered with plastic wrap and stored in the refrigerator as soon as possible.
  Other Names: Fresh lime (Citrus aurantifolia)

SUMMARY:
The purpose of this study is to determine whether fresh lime alone is effective for smoking cessation.

DETAILED DESCRIPTION:
Smoking is the major preventable cause of chronic medical diseases and death worldwide. Significant efforts led by World Health Organization (WHO) and several countries have been made to help current smokers to quit, particularly in the developing countries, where their smoking rates continued to rise. Clinical practice guidelines were therefore developed to guide all healthcare personnel in those countries to provide treatment for smokers. However, despite that, only a small number of smokers were able to quit successfully. A large number of smokers who are poor and heavily addicted to nicotine remain and have no access to any effective smoking cessation aids. Although there are several effective medications available for smoking cessation nowadays, the high price of them completely keeps poor smokers away from using them. Alternative and cheaper smoking cessation aids are therefore necessary. During the past decade, certain herbal remedies have been introduced in smoking cessation in Thailand. One of them that have been used widely without any supporting evidence is the fresh lime (Citrus aurantifolia), the well-known native citrus to Southeast Asia. It is anecdotally claimed to be effective and safe in smoking cessation. The present study was designed to determine the efficacy and safety of fresh lime as a smoking cessation aid compared with those of nicotine gum.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Smoked regularly at least one year prior to study entry
* Had the desire to quit smoking
* Signed informed consent

Exclusion Criteria:

* Having current dental problems
* Active peptic ulcer disease
* Psychiatric disorders
* Citrus allergy
* Pregnancy
* Use of illicit drugs
* Participation in another clinical trial and/or using any first-line smoking cessation aids within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
continuous abstinence rate (CAR) of lime group and gum group | week 12
  CAR from week 9 through week 12 of treatment was defined as proportion of participants who self-reported having refrained from smoking any tobacco products and confirmed by exhaled CO concentration of 10 ppm or less at all previous measurement points between week 9 and week 12 of treatment.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events on each group | week 12
  All adverse events related to the use of nicotine gum and fresh lime during the 12-week treatment were measured as number and percent of participants in each group.
7-day point prevalence abstinence (PAR) of lime and gum groups | week 4
  Point prevalence abstinence rate (PAR), which was defined as percentage of participants who were able to abstain from smoking any tobacco products during the preceding week, was evaluated at week 4, 8, 12 and 24.
7-day point prevalence abstinence (PAR) of lime and gum groups | week 8
  Point prevalence abstinence rate (PAR), which was defined as percentage of participants who were able to abstain from smoking any tobacco products during the preceding week, was evaluated at week 4, 8, 12 and 24.
7-day point prevalence abstinence (PAR) of lime and gum groups | week 12
  Point prevalence abstinence rate (PAR), which was defined as percentage of participants who were able to abstain from smoking any tobacco products during the preceding week, was evaluated at week 4, 8, 12 and 24.
continuous abstinence rates of the lime and gum groups | week 24
  CAR from week 9 through week 24 of the study was defined as proportion of participants who self-reported having refrained from smoking any tobacco products and confirmed by exhaled CO concentration of 10 ppm or less at all previous measurement points between week 9 and week 24.
intensity of craving using 100-mm VAS score | week 2
  Intensity of cravings after morning awakening among smokers in both groups were recorded on the day of clinic visits at week 2, 4, 8, 12, and 24 of the study using 100-mm visual analogue scale (VAS). Mean scores of those in the lime and gum groups was calculated and compared.
intensity of craving using 100-mm VAS score | week 4
  Intensity of cravings after morning awakening among smokers in both groups were recorded on the day of clinic visits at week 2, 4, 8, 12, and 24 of the study using 100-mm visual analogue scale (VAS). Mean scores of those in the lime and gum groups was calculated and compared.
intensity of craving using 100-mm VAS score | week 8
  Intensity of cravings after morning awakening among smokers in both groups were recorded on the day of clinic visits at week 2, 4, 8, 12, and 24 of the study using 100-mm visual analogue scale (VAS). Mean scores of those in the lime and gum groups was calculated and compared.
intensity of craving using 100-mm VAS score | week 12
  Intensity of cravings after morning awakening among smokers in both groups were recorded on the day of clinic visits at week 2, 4, 8, 12, and 24 of the study using 100-mm visual analogue scale (VAS). Mean scores of those in the lime and gum groups was calculated and compared.
intensity of craving using 100-mm VAS score | week 24
  Intensity of cravings after morning awakening among smokers in both groups were recorded on the day of clinic visits at week 2, 4, 8, 12, and 24 of the study using 100-mm visual analogue scale (VAS). Mean scores of those in the lime and gum groups was calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Suthat Rungruanghiranya, MD, Principal Investigator — Faculty of Medicine, Srinakharinwirot University
Locations (1):
- Panyananthaphikkhu Chonprathan Medical Center, Ban Plak Raet, Nondhaburi, Thailand

REFERENCES:
- [Result] Rungruanghiranya S, Ekpanyaskul C, Hattapornsawan Y, Tundulawessa Y. Effect of nicotine polyestex gum on smoking cessation and quality of life. J Med Assoc Thai. 2008 Nov;91(11):1656-62. PMID 19127785
- [Result] Lykkesfeldt J, Prieme H, Loft S, Poulsen HE. Effect of smoking cessation on plasma ascorbic acid concentration. BMJ. 1996 Jul 13;313(7049):91. doi: 10.1136/bmj.313.7049.91. No abstract available. PMID 8688760
- [Result] Levin ED, Behm F, Carnahan E, LeClair R, Shipley R, Rose JE. Clinical trials using ascorbic acid aerosol to aid smoking cessation. Drug Alcohol Depend. 1993 Oct;33(3):211-23. doi: 10.1016/0376-8716(93)90108-3. PMID 8261886